CLINICAL TRIAL: NCT01413035
Title: Safety/Efficacy Assessed Study on Transplantation Therapy Using Human Umbilical Cord/Placenta-derived Mesenchymal Stem Cells for Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy Study of Umbilical Cord/Placenta-Derived Mesenchymal Stem Cells to Treat Type 2 Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Chengyun Zheng, Department of Hematology of the 2nd Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: diabetes
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Diabetes Medicines: Oral Hypoglycemic Drugs and Insulins.; Umbilical Cord/placenta-Derived MSC; Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MSC and the oral hypoglycemic drugs (Experimental): 1.0E+6 MSC/kg, IV drop and repeat to apply in Day 90 if the effect of MSC is better. At the same time, patient continues to apply the former oral hypoglycemic drugs, such as Dimethylbiguanide, Glurenorm and Acarbose, et al. and regulates the dosage for 1 year.
  Interventions: Biological: MSC
- MSC and insulins (Experimental): 1.0E+6 MSC/kg, IV drop and repeat to apply in Day 90 if the effect of MSC is better. At the same time, patient continues to apply the former insulins and regulates the dosage for 1 year.
  Interventions: Biological: MSC
- MSC and the combination of drugs and insulins (Experimental): 1.0E+6 MSC/kg, IV drop and repeat to apply in Day 90 if the effect of MSC is better. At the same time, patient continues to apply the former combination of the oral hypoglycemic drugs and insulins and regulates the dosage for 1 year.
  Interventions: Biological: MSC

INTERVENTIONS:
Biological: MSC — 1.0E+6 MSC/kg, IV drop in Day 0 and repeat to apply in Day 90 if the effect of MSC is better.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells (MSCs) derived from human umbilical cord/placenta at a dose of 1.0E+6 MSC/kg for type 2 diabetes.

DETAILED DESCRIPTION:
1. Intervention Details: Biological: umbilical cord/placenta-derived mesenchymal stem cells; Drug: 1. Oral Hypoglycemic Drugs, such as Dimethylbiguanide, Glurenorm and Acarbose, et al. 2. Insulins.

1. 1st transplantation: after finishing all required examines according to protocol in Day 0, umbilical cord/placenta-derived MSCs are transplanted intravenously.
2. 2nd transplantation: after finishing all required examines in Day 90, umbilical cord/placenta-derived-MSCs are transplanted intravenously if the effects of MSC are better than that before.
3. At the same time, patients continue taking the oral hypoglycemic drugs, insulins or the combination of the oral hypoglycemic drugs and insulins which the patients have taken for controlling the higher blood sugar from Day 0 for 1 year. But the dose of the oral hypoglycemic drugs and insulins should be regulated according to the level of blood sugar.

2. Detailed Description:

1. To evaluate the feasibility and safety of transplantation treatment using umbilical cord/placenta-derived mesenchymal stem cells in patients with type 2 diabetes mellitus undergoing the oral hypoglycemic drugs, insulins or the combination of the oral hypoglycemic drugs and insulins.
2. To assess efficacy of transplantation treatment using umbilical cord/placenta-derived mesenchymal stem cells in patients with type 2 diabetes mellitus undergoing the oral hypoglycemic drugs, insulins or the combination of the oral hypoglycemic drugs and insulins.
3. This study will last 2 to 3 years. Participants will be randomly assigned to receive either MSC transplant and the oral hypoglycemic drugs or MSC transplant and insulins or MSC transplant and the combination of the oral hypoglycemic drugs and insulins (experimental group) or the oral hypoglycemic drugs or insulins or the combination of the oral hypoglycemic drugs and insulins (control group). Patients will undergo MSC transplant at the start of the study on Day 0 and take the oral hypoglycemic drugs, insulins or the combination of the oral hypoglycemic drugs and insulins for 1 year. As control, some patients take the oral hypoglycemic drugs, insulins or the combination of the oral hypoglycemic drugs and insulins for 1 year. At the same time, the dose of the oral hypoglycemic drugs and insulins should be regulated according to the level of blood sugar. After 3 months, patients will receive the second MSC transplantation. After six and twelve months from the first transplantation, patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Free will taking part in the study and ability to provide written informed consent
* Type 2 diabetes mellitus (as guideline WHO, 1999)
* Age 18-80 years old, Male/Female
* 19≤Body mass index (BMI)≤30㎏/㎡
* Fast blood glucose (FBG)≥7.0 mmol/L, and HbAc1≥7％
* Intravenous insulin tolerance test（ITT）indicate patient being insulin resistance
* Not pregnant or nursing
* No moderate or sever organ dysfunction: Ejection fraction>45%; Creatinine <176 mmol/L
* No active severe viral or fungus infection

Exclusion Criteria:

* Severe concurrent medical condition (e.g., serious heart disease, lung disease, or hematopoietic dysfunction, or liver dysfunction, or kidney dysfunction)
* Active infection requiring treatment
* Unexplained febrile illness
* Known immunosuppressive disease, e.g. HIV infection, or hepatitis B or C infection
* Psychiatric condition that would limit informed consent
* Patient has enrolled another clinical trial study within last 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
To assess efficacy of transplantation treatment using umbilical cord/placenta-derived mesenchymal stem cells in patients with type 2 diabetes mellitus | 1 year
  To assess efficacy of MSC through comparing the change of ITT, Hemoglobin A1c, FBG, PBG, C-peptide levels and T cell subsets with that of baseline.
  1. The change of insulin resistance index(ITT) compared with baseline.
  2. Rate of reducing exogenous insulin requirement compared with baseline.
  3. The change of Fast blood glucose (FBG) and Postmeal blood glucose (PBG) compared with baseline.
  4. A reduction of ≥1% in HbA1c compared with baseline.
  5. The change of C-peptide levels compared with baseline.
  6. The change of T cell subsets compared with baseline.

SECONDARY OUTCOMES:
To evaluate the incidence and severity of adverse events of transplantation treatment using umbilical cord/placenta-derived mesenchymal stem cells in patients with type 2 diabetes mellitus | 1 year
  To evaluate if there have occured the adverse everts such as fever, allergy, et al. and their severity.

CONTACTS AND LOCATIONS:
Overall Officials: chengyun zheng, Ph. D, Principal Investigator — Department of Hematology of The 2nd Hospital of Shandong University
Locations (1):
- Department of Hematology of the 2nd Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Kong D, Zhuang X, Wang D, Qu H, Jiang Y, Li X, Wu W, Xiao J, Liu X, Liu J, Li A, Wang J, Dou A, Wang Y, Sun J, Lv H, Zhang G, Zhang X, Chen S, Ni Y, Zheng C. Umbilical cord mesenchymal stem cell transfusion ameliorated hyperglycemia in patients with type 2 diabetes mellitus. Clin Lab. 2014;60(12):1969-76. doi: 10.7754/clin.lab.2014.140305. PMID 25651730